CLINICAL TRIAL: NCT04080414
Title: Home-based High-intensity Interval Training to Improve Colorectal Cancer Survivorship: Feasibility and Relationship With Novel Surrogate Biomarkers of Colorectal Cancer Recurrence
Brief Title: Home-based HIIT to Improve CRC Survivorship: Feasibility and Relationship With Novel Surrogate Biomarkers of CRC Recurrence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Adriana Coletta, Assistant Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 122238
Record Dates: First submitted 2019-08-12; First posted 2019-09-06 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Colorectal Cancer; Colorectal Neoplasms; Colorectal Carcinoma; Colonic Neoplasms; Colonic Cancer; Rectal Neoplasms; Rectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based high-intensity interval training (Experimental)
  Interventions: Behavioral: Home-based high-intensity interval training
- Home-based moderate-intensity continuous exercise (Active Comparator)
  Interventions: Behavioral: Home-based moderate-intensity continuous exercise

INTERVENTIONS:
Behavioral: Home-based high-intensity interval training — Participants will be instructed to complete four, high-intensity interval training workouts per week at home, for the duration of the 12-week trial. Participants will be provided with detailed instructions on how to complete each workout.
  Arms: Home-based high-intensity interval training
Behavioral: Home-based moderate-intensity continuous exercise — Participants will be instructed to complete five, moderate-intensity continuous exercise workouts per week at home, for the duration of the 12-week trial. Participants will be provided with detailed instructions on how to complete each workout.
  Arms: Home-based moderate-intensity continuous exercise

SUMMARY:
This 12-week, exercise study will assess the feasibility of a home-based high-intensity interval training (HIIT) program among colorectal cancer survivors and explore the impact of home-based HIIT compared to a standard home-based moderate-intensity continuous aerobic exercise program on physical outcomes linked with survival from colorectal cancer and surrogate blood markers of colorectal cancer recurrence.

HIIT is a type of aerobic exercise that includes short bursts (i.e. 1-4 minutes) of vigorous exercise followed by longer periods of moderate to lower intensity exercise (i.e. 1-10 minutes). Participants in this study will be randomly assigned into a personalized home based exercise program - either high-intensity interval training (HIIT) or moderate-intensity continuous aerobic exercise (MICE).

This pilot study will provide us with preliminary evidence for a larger trial aimed to compare the effectiveness of these two different types of home-based exercise programs on physical outcomes linked with survival, quality of life, and surrogate blood markers of colorectal cancer recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are no more than five years post resection and/or adjuvant therapy for stage II-III Colorectal cancer (CRC).
2. Age 19-75 years old.
3. Engaging in less than 90 minutes per week of structured moderate- or vigorous-intensity aerobic exercise in the past three months
4. No known cardiovascular, metabolic or renal disease, and no signs/symptoms suggestive of cardiovascular, metabolic, or renal disease.
5. Must be able to read, speak and understand English
6. Willing to complete two assessment sessions (at baseline and 12 weeks).
7. Willing to engage in moderate- or vigorous-intensity aerobic exercise at home and use mobile health technology to track exercise adherence to the exercise prescription.
8. Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.
9. Have regular access to a smart phone and willing to download a free application for device tracking

Exclusion Criteria:

1. Functional limitations requiring a walker, scooter, or wheelchair.
2. Clinically evident recurrent disease.
3. Resting blood pressure ≥140/90 at the time of baseline testing.
4. No access to smart phone and/or not willing download the device app

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-08-02 (Actual); Primary Completion 2021-02-12 (Actual); Study Completion 2021-02-12 (Actual)

PRIMARY OUTCOMES:
Feasibility of home-based high-intensity interval training among colorectal cancer survivors | 12 weeks
  Feasibility will be assessed by adherence to the home-based high-intensity interval training protocol, which is defined at the participant level as completing ≥70% of workouts consistent with the exercise prescription. The intervention will be considered feasible if ≥75% of participants meet or exceed the 70% criterion.

CONTACTS AND LOCATIONS:
Overall Officials: Adriana M Coletta, PhD, Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - Intermountain Medical Center, Murray, Utah
  - Huntsman Cancer Institute at the University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No